CLINICAL TRIAL: NCT05475223
Title: End Tidal Carbon Monoxide (ETCO) : A Tool to Aid Identification of Neonatal Hemolysis
Brief Title: End Tidal Carbon Monoxide (ETCO): - A Tool to Aid Identification of Neonatal Hemolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jyotirbala Ruparel, MD, Medical Director, HRIF, CSMC, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00000491
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: End Tidal Carbon Monoxide Excretion as a Diagnostic Tool for Hemolysis in the Newborn; Neonatal Jaundice; End Tidal Carbon Monoxide
Keywords: Neonatal Hemolysis; Neonatal Jaundice; ETCO; End Tidal Carbon Monoxide
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: Retrospective review of subjects for Standard of Care for Neonatal jaundice diagnosis and management (SOC) will be compared with a prospective group of subjects with Standard of care for Neonatal jaundice for diagnosis and management + End Tidal Carbon Monoxide management (ETCO)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective (Other): Standard of Care for Diagnosis and management of neonatal jaundice + End Tidal Carbon Monoxide measurement value
  Interventions: Diagnostic Test: End Tidal Carbon Monoxide Value

INTERVENTIONS:
Diagnostic Test: End Tidal Carbon Monoxide Value — A noninvasive ETCO value will be obtained by inserting a soft silicon cannula placed in the baby's nostril for a few minutes to measure exhaled end tidal carbon monoxide; a value corrected for ambient ETCO value will be recorded.

SUMMARY:
The purpose of this study is to evaluate if adding a noninvasive testing of End Tidal Carbon Monoxide with a FDA approved device will help improve management of jaundice in the Neonates by reducing the number of lab draws, Coombs tests and optimizing the number of phototherapy hours in Neonates who need it.

Eligible subjects will be Term and healthy late preterm newborns born at Cedars-Sinai Medical Center and admitted to well baby nursery from November 2020 onwards.

The primary procedure of measuring an End-Tidal Carbon monoxide in a Newborn is going to be with a soft cannula applied to the Newborn's nose for a few minutes. The whole procedure will take about 15+ 5 minutes.

Subject participation will last approximately 6 months and all subjects will be followed up with one phone call at about 2-4 weeks of age.

Adding ETCO testing to current standard of care might reduce the number of lab draws in a newborn and potentially reduce costs by optimizing the number of phototherapy hours in a Newborn who needs it. Cedars- Sinai Medical Center will not be billing the patients for the End-Tidal Carbon Monoxide measurement for this study.

DETAILED DESCRIPTION:
The purpose the research is:

* Whether near simultaneous measurements of Total Serum bilirubin (Tsb) & End-Tidal Carbon Monoxide (End-Tidal Carbon monoxide as a function of bilirubin) will help identify hyperbilirubinemia accurately and easily This has been shown in a single center study.
* Whether near simultaneous measurement of Total serum bilirubin & End Tidal Carbon Monoxide is more accurate and less costly in overall management of Neonatal Hyperbilirubinemia Eligible infants would be male or female with GA > 35 weeks and BW > 2000, post natal age 6 hours to < 6 days of age and meets any one of the following criteria
* Due for an early discharge
* Has a Transcutaneous bilirubin or a Total serum bilirubin on or > the 75th % of Bhutani hyperbilirubinemia nomogram
* Has 2 or more risk factors for neonatal jaundice as specified in the protocol
* The study includes 388 patients in each arm - ~ 776 total newborn admissions
* The total study duration is: 6 months Methods: a retrospective group (Standard of Care) will be compared with a prospective Group (Standard of care + End-Tidal Carbon monoxide). Informed Consent will be obtained before the subject is recruited in the prospective group.

A phone call will be made to each subject in the prospective group at 2-4 weeks of age post birth hospitalization. This is a minimally risk study.

ELIGIBILITY:
Inclusion Criteria:

* male or female with GA > 35 weeks and BW > 2000, post natal age 6 hours to < 6 days of age and meets any one of the following criteria

  * Due for an early discharge
  * Has a TcB or Tsb on or > the 75th % of Bhutani hyperbilirubinemia nomogram
  * Has 2 or more risk factors for neonatal jaundice as specified in the protocol

Exclusion Criteria:

* babies requiring any kind of respiratory support (O2, CPAP or assisted ventilation) has severe or life threatening congenital anomalies, weighed less than 2000 gms and if their mother has a known history of smoking during 3rd trimester of pregnancy. Also in addition nasal mucosal abrasion or nasal mucosal abnormalities will be excluded.

Ages: 35 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Estimated)
Dates: Start 2022-07-29 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in usage of Coombs Test and other Labs Ordered for hemolysis in Neonatal Jaundice | 6 months
  We expect a projected change of 10-15% in Coombs Test usage for neonatal jaundice and mean difference of 1 in other labs ordered for hemolysis in neonatal jaundice

SECONDARY OUTCOMES:
Adding ETCO to diagnostic procedures for hemolysis in neonatal jaundice will help optimize phototherapy | 6 months
  On average on readmission at Cedars- Sinai Medical Center a newborn gets 36 +/-10 hours of phototherapy and on birth admission some babies are getting 6 +/- 12 hours of phototherapy. ETCO (End tidal carbon monoxide value) used a function of Total serum bilirubin will help optimize the number of hours of phototherapy.
Recording of nursing time to perform the test | 6 months
  The time taken by medical personnel to perform and record results will be recorded

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Background] Tidmarsh GF, Wong RJ, Stevenson DK. End-tidal carbon monoxide and hemolysis. J Perinatol. 2014 Aug;34(8):577-81. doi: 10.1038/jp.2014.66. Epub 2014 Apr 17. PMID 24743136
- [Background] Bhutani VK, Srinivas S, Castillo Cuadrado ME, Aby JL, Wong RJ, Stevenson DK. Identification of neonatal haemolysis: an approach to predischarge management of neonatal hyperbilirubinemia. Acta Paediatr. 2016 May;105(5):e189-94. doi: 10.1111/apa.13341. Epub 2016 Feb 29. PMID 26802319
- [Background] Christensen RD, Malleske DT, Lambert DK, Baer VL, Prchal JT, Denson LE, Gerday E, Weaver Lewis KA, Shepherd JG. Measuring End-Tidal Carbon Monoxide of Jaundiced Neonates in the Birth Hospital to Identify Those with Hemolysis. Neonatology. 2016;109(1):1-5. doi: 10.1159/000438482. Epub 2015 Sep 23. PMID 26394287
- [Background] Bhutani VK, Johnson L, Sivieri EM. Predictive ability of a predischarge hour-specific serum bilirubin for subsequent significant hyperbilirubinemia in healthy term and near-term newborns. Pediatrics. 1999 Jan;103(1):6-14. doi: 10.1542/peds.103.1.6. PMID 9917432
- [Background] Kuzniewicz M, Newman TB. Interaction of hemolysis and hyperbilirubinemia on neurodevelopmental outcomes in the collaborative perinatal project. Pediatrics. 2009 Mar;123(3):1045-50. doi: 10.1542/peds.2007-3413. PMID 19255038